# The Influence of Cognitive Behavioral Therapy on Fatigue, Cognition and Inflammatory Biomarkers in Multiple Sclerosis Patients: Single Blinded Randomized Controlled Trial

**Protocol** 

# By

## ENGY BADRELDIN SALEH MOUSTAFA

PhD., Lecturer in Faculty of Physical Therapy
Department for Neuromuscular Disorders & its Surgery
Cairo University

### **SUPERVISORS**

### Prof. Dr. Moshera Hassan Darwish

Professor of Physical Therapy for Neuromuscular Disorder & its Surgery Faculty of Physical Therapy Cairo University

> Faculty of Physical Therapy Cairo University 2020

# **Ethical Committee Approval Number**



# Appendix (I)

### SAMPLE CONSENT FORM

I am....freely and voluntarily consent to participate in a research program under the direction of M.Sc. Ahmed shawky.

A thorough description of the procedure has been explained and I understand that I may withdraw my consent and discontinue participation in this research at any time without prejudice to me.

Date Participant

23/12/2020